CLINICAL TRIAL: NCT02838199
Title: Prospective, Open Label, Multicenter, Dual Arm, Randomized Trial of TRANscatheter or SurgIcal Aortic Valve ReplacemenT in All-Comers With Severe Aortic Valve Stenosis
Brief Title: TRANscatheter or SurgIcal Aortic Valve ReplacemenT in All-Comers With Severe Aortic Valve Stenosis
Acronym: TRANSIT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-16
Record Dates: First submitted 2016-07-06; First posted 2016-07-20 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter aortic valve replacement; TAVR; TAVI; SAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAVR (Experimental): Transcatheter aortic valve replacement with SAPIEN 3
  Interventions: Device: SAPIEN 3
- SAVR (Active Comparator): Surgical aortic valve replacement
  Interventions: Procedure: SAVR

INTERVENTIONS:
Device: SAPIEN 3
  Arms: TAVR
Procedure: SAVR
  Arms: SAVR

SUMMARY:
The purpose of this study is to determine that Transcatheter aortic valve replacement (TAVR) with SAPIEN 3 is superior to traditional surgical aortic valve replacement(SAVR) with bio-prosthesis regarding the rate of all-cause mortality at 1 year in patients with symptomatic severe aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age must be at least 19 and less than 75 years old
* Severe aortic valve stenosis with echocardiographically derived criteria: mean gradient > 40mmHg or jet velocity greater than 4.0 m/s AND an initial aortic valve area (AVA) of ≤ 0.8 cm2. Echocardiogram must be within 3 months of the date of the procedure
* Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA class II or greater.
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Life expectancy <1 year due to medical illness
* Suspected Malignancy
* Inoperability evaluated by surgeon
* Concomitant severe coronary artery disease not amenable for percutaneous coronary intervention
* Concomitant severe mitral valve or significant aorta disease requiring surgery
* Active bacterial endocarditis within 6 months of procedure
* Leukopenia (WBC<3000 cell/mL), acute anemia (Hgb<8g/dL), thrombocytopenia (platelet < 50000 cell/mL)
* Intracardiac thrombus
* A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
* Native aortic annulus size < 18 mm or > 25 mm as measured by echocardiogram.
* Expectation that patient will not improve despite treatment of aortic stenosis
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2020-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
event rate of all-cause mortality | 1 year

SECONDARY OUTCOMES:
event rate of cardiovascular mortality | 30 days or hospital discharge, whichever is longer
event rate of cardiovascular mortality | 31 days to the 1 year
event rate of myocardial Infarction | 30 days or hospital discharge, whichever is longer
event rate of myocardial Infarction | 31 days to the 1 year
event rate of all Stroke and transient ischemic attack | 30 days or hospital discharge, whichever is longer
event rate of all Stroke and transient ischemic attack | 31 days to the 1 year
event rate of bleeding | 30 days or hospital discharge, whichever is longer
event rate of bleeding | 31 days to the 1 year
event rate of vascular access site and access-related complication | 30 days or hospital discharge, whichever is longer
event rate of vascular access site and access-related complication | 31 days to the 1 year
event rate of acute kidney injury | 30 days or hospital discharge, whichever is longer
event rate of acute kidney injury | 31 days to the 1 year
event rate of permanent pacemaker insertion | 30 days or hospital discharge, whichever is longer
event rate of permanent pacemaker insertion | 31 days to the 1 year
event rate of other TAVR-related complication | 30 days or hospital discharge, whichever is longer
  Conversion to open surgery Coronary obstruction Mitral valve apparatus damage or dysfunction Cardiac tamponade Endocarditis Valve thrombosis Valve malpositioning TAV-in-TAV deployment
event rate of other TAVR-related complication | 31 days to the 1 year
  Conversion to open surgery Coronary obstruction Mitral valve apparatus damage or dysfunction Cardiac tamponade Endocarditis Valve thrombosis Valve malpositioning TAV-in-TAV deployment
event rate of prosthetic valve dysfunction | 30 days or hospital discharge, whichever is longer
  Prosthetic aortic valve stenosis Prosthesis-patient mismatch Prosthetic aortic valve regurgitation
event rate of prosthetic valve dysfunction | 31 days to the 1 year
  Prosthetic aortic valve stenosis Prosthesis-patient mismatch Prosthetic aortic valve regurgitation
event rate of composite event for device success, early safety, clinical efficacy | 30 days or hospital discharge, whichever is longer
  Number of cases with following events ;
  A. Device success
  or
  B. Early safety (At 30 days):
  All-cause mortality, all stroke, life threatening bleeding, acute kidney injury, coronary obstruction requiring intervention, major vascular complication, valve-related dysfunction requiring repeat procedure.
  or
  C. Clinical efficacy (After 30 days):
  All-cause mortality, all stroke, requiring hospitalization for valve-related symptoms or worsening congestive heart failure, NYHA class III or IV, valve related dysfunction.
event rate of composite event for device success, early safety, clinical efficacy | 31 days to the 1 year
  Number of cases with following events ;
  A. Device success
  or
  B. Early safety (At 30 days):
  All-cause mortality, all stroke, life threatening bleeding, acute kidney injury, coronary obstruction requiring intervention, major vascular complication, valve-related dysfunction requiring repeat procedure.
  or
  C. Clinical efficacy (After 30 days):
  All-cause mortality, all stroke, requiring hospitalization for valve-related symptoms or worsening congestive heart failure, NYHA class III or IV, valve related dysfunction.
event rate of structural valve deterioration | 30 days or hospital discharge, whichever is longer
event rate of structural valve deterioration | 31 days to the 1 year
NYHA (New York Heart Association Functional Classification) | 30days and 1 year
Valve area | 30days and 1 year
  Aortic valve area (AVA) measured by 2D-transthoracic echocardiography using the continuity equation.
event rate of free from atrial fibrillation | 30days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suck-jung Choo, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided